CLINICAL TRIAL: NCT05729659
Title: The Effect of Sideritis Scardica (SidTea+) Extract Supplementation on Health and Oxidative Stress Biomarkers in Healthy Individuals
Brief Title: Sideritis Supplementation, Oxidative Stress and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Z. Jamurtas, Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UTH-DPESS_Sideritis
Record Dates: First submitted 2023-01-16; First posted 2023-02-15 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Oxidative Stress; Lipidemia
Keywords: Sideritis; Extract; Antioxidants; Oxidative stress; Health
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sideritis Scardica (SidTea+) extract (Experimental): Sideritis Scardica (SidTea+) extract will be administered to participants in this arm.
  Interventions: Dietary Supplement: Sideritis Scardica (SidTea+) extract supplementation
- Placebo (Placebo Comparator): Placebo will be administered to participants in this arm.
  Interventions: Dietary Supplement: Placebo supplementation

INTERVENTIONS:
Dietary Supplement: Sideritis Scardica (SidTea+) extract supplementation — 1500 mg of Sideritis Scardica (SidTea+) extract per day, divided into 3 equal doses of 500 mg (every 8 hours) for a total duration of 1 month
  Arms: Sideritis Scardica (SidTea+) extract
Dietary Supplement: Placebo supplementation — 1500 mg of placebo per day, divided into 3 equal doses of 500 mg (every 8 hours) for a total duration of 1 month
  Arms: Placebo

SUMMARY:
The aim of the present clinical study is to estimate the efficacy of a Sideritis Scardica extract (SidTea+), derived from the Greek mountain Taygetos, in regulating antioxidant and health biomarkers in healthy adults.

DETAILED DESCRIPTION:
Introduction: The mountain tea of genus Sideritis has more than 150 species, which are mainly distributed in the Mediterranean area. In the literature, extensive reference is made to the secondary metabolites of Sideritis, the main ones of which are terpenoids (i.e., iridoids and kauranes) and phenolic derivatives (i.e., flavonoids, phenolic acids, phenylethanoid glycosides). Polyphenols exhibit a wide range of biological activities, such as anti-atherogenic, anti-cancer, anti-mutagenic, anti-inflammatory and antimicrobial properties. Among phenolic derivatives, major significance is given to flavonoids, due to their antioxidant, anti-inflammatory, antibacterial, antiviral and anti-allergic properties in various pathologies. Flavonoids mainly act as antioxidants, inhibiting free radical-induced cytotoxicity and lipid peroxidation. Moreover, these compounds are known to inhibit tumor growth and proliferation and act as weak agonists or antagonists of estrogens by regulating endogenous hormonal activity. In these ways, they can protect against chronic diseases such as atherosclerosis and cancer and regulate menopausal symptoms.

Purpose: This study aims to investigate the effect of a Sideritis Scardica extract (SidTea+) supplement from the Greek mountain Taygetos on health and oxidative stress indicators in healthy individuals. The results of the present investigation will help to elucidate the effects of an extract derived from a plant product on markers of health and oxidative stress in apparently healthy individuals.

Methodology: 30 healthy individuals will be enrolled in the study. Participants will give their informed consent after they will be informed about the purposes, procedures, risks and benefits associated with the study. Participants will be randomly allocated to either a Sideritis spp or a placebo supplementation group and they will consume 1500 mg/day of Sideritis or placebo, distributed in three equal doses (every 8 hours) for one month. At baseline and post-intervention, volunteers will be assessed for their anthropometric profile, muscle function and cardiorespiratory capacity and will provide a resting blood sample for the assessment of oxidative stress and health biomarkers. Participants will be asked to record their diet for 3 days prior to the study and they will be asked to follow the same dietary pattern for 3 days before the post-intervention assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Individuals aged 18-65 years

Exclusion Criteria:

* Musculoskeletal injury
* Dietary supplements
* Medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in glutathione concentration | Change from baseline to 1 month
  Glutathione concentration will be analyzed in erythrocytes
Change in catalase activity | Change from baseline to 1 month
  Catalase activity will be analyzed in erythrocytes
Change in total antioxidant capacity | Change from baseline to 1 month
  Total antioxidant capacity will be analyzed in serum
Change in thiobarbituric acid reactive substances concentration | Change from baseline to 1 month
  Thiobarbituric acid reactive substances concentration will be analyzed in plasma
Change in protein carbonyls concentration | Change from baseline to 1 month
  Protein carbonyls will be analyzed in plasma
Change in glucose concentration | Change from baseline to 1 month
  Glucose concentration will be analyzed in plasma
Change in cholesterol concentration | Change from baseline to 1 month
  Cholesterol concentration will be analyzed in plasma
Change in triglycerides concentration | Change from baseline to 1 month
  triglycerides concentration will be analyzed in plasma
Change in high-density lipoprotein concentration | Change from baseline to 1 month
  High-density lipoprotein concentration will be analyzed in plasma
Change in bilirubin concentration | Change from baseline to 1 month
  Bilirubin concentration will be analyzed in plasma
Change in lactate dehydrogenase concentration | Change from baseline to 1 month
  Lactate dehydrogenase concentration will be analyzed in plasma
Change in serum glutamic-oxaloacetic transaminase concentration | Change from baseline to 1 month
  Serum glutamic-oxaloacetic transaminase will be analyzed in serum
Change in gamma-glutamyl transpeptidase concentration | Change from baseline to 1 month
  Gamma-glutamyl transpeptidase concentration will be analyzed in serum
Change in creatinine concentration | Change from baseline to 1 month
  Creatinine concentration will be analyzed in serum
Change in uric acid concentration | Change from baseline to 1 month
  Uric acid concentration will be analyzed in serum

SECONDARY OUTCOMES:
Change in handgrip strength | Change from baseline to 1 month
  Handgrip strength will be measured using a hand dynamometer
Change in estimated maximal oxygen consumption (eVO2max) | Change from baseline to 1 month
  eVO2max will be measured using an automated open-circuit spirometer
Change in body weight | Change from baseline to 1 month
  Body weight will be measured using a digital scale
Change in body fat | Change from baseline to 1 month
  Body fat will be measured by bioelectrical impedance analysis
Change in resting heart rate | Change from baseline to 1 month
  Resting heart rate will be measured using a heart rate sensor
Change in diastolic and systolic blood pressure | Change from baseline to 1 month
  Diastolic and systolic blood pressure will be measured using a manual sphygmomanometer
Change in waist and hip circumference | Change from baseline to 1 month
  Waist and hip circumference will be assessed using a tape measure
Change in complete blood count | Change from baseline to 1 month
  White blood cells, lymphocytes, monocytes, granulocytes, red blood cells and platelets will be analyzed in whole blood using an automated blood chemistry analyzer
Dietary macro-nutrient analysis | Baseline
  Protein, carbohydrate and fat dietary intake will be measured using diet recalls (food questionnaires)
Dietary micro-nutrient analysis | Baseline
  Vitamin C, vitamin E, zinc, methionine and cysteine dietary intake will be analyzed using diet recalls (food questionnaires)
Physical activity level | Baseline
  Low, moderate and vigorous physical activity will be assessed by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Z. Jamurtas, Professor, Study Director — University of Thessaly; Konstantinos Papanikolaou, PhD, Principal Investigator — University of Thessaly
Locations (1):
- Exercise Biochemistry, Physiology and Nutrition Laboratory, Department of Physical Education and Sport Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsaknis J, Lalas S. Extraction and identification of natural antioxidant from Sideritis euboea (mountain tea). J Agric Food Chem. 2005 Aug 10;53(16):6375-81. doi: 10.1021/jf0479261. PMID 16076121
- [Background] Gabrieli CN, Kefalas PG, Kokkalou EL. Antioxidant activity of flavonoids from Sideritis raeseri. J Ethnopharmacol. 2005 Jan 15;96(3):423-8. doi: 10.1016/j.jep.2004.09.031. Epub 2004 Nov 6. PMID 15619561
- [Background] Yao LH, Jiang YM, Shi J, Tomas-Barberan FA, Datta N, Singanusong R, Chen SS. Flavonoids in food and their health benefits. Plant Foods Hum Nutr. 2004 Summer;59(3):113-22. doi: 10.1007/s11130-004-0049-7. PMID 15678717